CLINICAL TRIAL: NCT02179450
Title: Pilot Study Assessing Cognitive Function and Emotional Possessing in Patients With Bilateral Facial Palsy
Brief Title: Cognitive Function and Emotional Possessing in Bilateral Facial Palsy
Status: Completed | Type: Observational
Sponsor: Kirsten Elwischger, MD (Other)
Responsible Party: Sponsor-Investigator, Kirsten Elwischger, MD, Dr. Kirsten Elwischger, Medical University of Vienna
Organization: Medical University of Vienna (Other)
Other Study IDs: Cognition_Facial palsy
Record Dates: First submitted 2012-12-31; First posted 2014-07-01 (Estimated); Last update posted 2014-07-01 (Estimated); Status verified 2014-06

CONDITIONS: Intelligence; Emotion

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Blepharospasm: Patients suffering from Blepharospasm
- Cervical Dystonia: Patients suffering from cervical dystonia
- Bilateral facial palsy: Patients suffering from bilateral facial palsy of inflammatory origin
- Healthy Control: Control subjects

SUMMARY:
Based on recent findings that botulinum toxin injections in the cranial muscles might reduce emotional processing (Havas 2011), an increasing number of popular newspaper tabloids are suggesting a negative effect on cognition. The underlying research articles address the "facial feedback hypothesis". The hypothesis indicates that expressive behaviour, including facial mimic expressions influences the subject's brain via feedback. (Alam 2008) Other systemic neurological diseases, e.g of inflammatory origin, may lead to temporary bilateral facial nerve palsy (BF). During recovery process, the palsy usually remits completely.

The effect of bilateral facial muscle palsy on cognition and emotional possessing has never been evaluated.

The results of this pilot study might provide new information about the effect bilateral facial palsy on emotional processing and cognition and the facial feedback hypothesis.

The aim of this controlled pilot study is to assess cognitive function and emotional processing in patients with bilateral facial palsy. In addition, differences in cognitive function and emotional processing in patients with different manifestations of dystonia should be evaluated.

According to the facial feedback theory, paralysed mimic muscles might alter emotional processing. Therefore, investigators compare patients with bilateral facial muscle palsy and healthy controls. Investigators expect no influence of facial muscle palsy on cognitive functions in any of the tested groups; the investigators expect a mild impairment of emotional processing only in the patients group with bilateral facial muscle palsy (BEB and BF). In addition, the investigators expect no difference in emotional processing in patients with different manifestations of dystonia (BEB and CD) at remission. There might be a slight difference of emotional processing in patients with different manifestations of dystonia (BEB and CD) at time of prominent facial palsy.

ELIGIBILITY:
Inclusion Criteria:

Patients:

* willing to participate in this pilot trial
* bilateral facial palsy
* age 18-80 years

Control:

* willing to participate in this pilot trial
* age,
* gender and
* education (duration of school attendance) matched
* and/or cervical dystonia

Exclusion Criteria:

* neurological or psychiatric comorbidity
* psychotropic drugs

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Two patient groups with bilateral facial palsy, 31 patients each (group A: BEB, , group C: BF), recruited from the Botulinum toxin outpatient's clinic and general outpatient's clinic of the Medical University of Vienna. Two control groups, 31 patients with CD, recruited from the Botulinum toxin outpatient's clinic of the Medical University of Vienna, and and 31 age-and education-matched HC, will perform neuropsychological testing of approximately 60 minutes duration at time of prominent facial palsy (baseline) and at remission (visit 1). HC age and education matched, will be tested twice.
  A total of 124 persons will be tested. All participants will sign an informed consent form. Group A: 31 BEB Group B: 31 CD Group C: 31 BF Group D: 31 HC
Sampling Method: Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2012-08; Primary Completion 2013-05 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
I-S-T-2000R- (intelligence-structure-test 2000R) | up to four weeks
  Test to evaluate Intelligence
  * Subtest "Matrixes"
  * Subtest "Analogies"

SECONDARY OUTCOMES:
Beck's depression-inventory-II | up to four weeks
  Evaluation of depression (BDI-II; Hautzinger et al., 2009)
Apathy Evaluation Scale | up to four weeks
  Evaluation of apathy (AES; Luecken et al., 2006)

CONTACTS AND LOCATIONS:
Overall Officials: Eduard Auff, Prof., MD, Principal Investigator — Department of Neurology, Medical University of Vienna
Locations (1):
- Department of Neurology, Medical University of Vienna, Vienna, Vienna, Austria

REFERENCES:
- [Background] Havas DA, Glenberg AM, Gutowski KA, Lucarelli MJ, Davidson RJ. Cosmetic use of botulinum toxin-a affects processing of emotional language. Psychol Sci. 2010 Jul;21(7):895-900. doi: 10.1177/0956797610374742. Epub 2010 Jun 14. PMID 20548056
- [Background] Alam M, Barrett KC, Hodapp RM, Arndt KA. Botulinum toxin and the facial feedback hypothesis: can looking better make you feel happier? J Am Acad Dermatol. 2008 Jun;58(6):1061-72. doi: 10.1016/j.jaad.2007.10.649. PMID 18485989
- [Background] Hennenlotter A, Dresel C, Castrop F, Ceballos-Baumann AO, Wohlschlager AM, Haslinger B. The link between facial feedback and neural activity within central circuitries of emotion--new insights from botulinum toxin-induced denervation of frown muscles. Cereb Cortex. 2009 Mar;19(3):537-42. doi: 10.1093/cercor/bhn104. Epub 2008 Jun 17. PMID 18562330
- [Derived] Platho-Elwischger K, Schmoeger M, Willinger U, Abdel-Aziz C, Algner J, Pretscherer S, Auff E, Kranz G, Turnbull O, Sycha T. Cognitive Performance After Facial Botulinum Toxin Treatment in a Cohort of Neurologic Patients: An Exploratory Study. Arch Phys Med Rehabil. 2022 Mar;103(3):402-408. doi: 10.1016/j.apmr.2021.08.007. Epub 2021 Sep 5. PMID 34496270